CLINICAL TRIAL: NCT02686905
Title: Effects of Vitamin Supplementation on Micronutrient Blood Values, Body Composition, Waist-to-hip Ratio and Fasting Blood Glucose After Bariatric Surgery
Brief Title: Vitamin Supplementation After Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: California State Polytechnic University, Pomona (Other)
Responsible Party: Principal Investigator, Rebecca McDorman, Graduate Student, California State Polytechnic University, Pomona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VitaBari Study
Record Dates: First submitted 2016-02-04; First posted 2016-02-22 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Complications of Bariatric Procedures; Avitaminosis
MeSH Terms: conditions — Avitaminosis | interventions — Iron; Transdermal Patch; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical vitamin patch (Experimental): Dietary Supplement: PatchMD Vitamin D3/Calcium Patch Dietary Supplement: PatchMD Multivitamin Patch Dietary Supplement: PatchMD B12 Energy Plus Patch
  Interventions: Dietary Supplement: PatchMD Vitamin D3/Calcium Patch; Dietary Supplement: PatchMD Multivitamin Patch; Dietary Supplement: PatchMD B12 Energy Plus Patch
- Oral vitamins (Experimental): Dietary Supplement: Chewable Multivitamin with Iron Dietary Supplement: Chewable Calcium Dietary Supplement: Quick Dissolve B12
  Interventions: Dietary Supplement: Chewable Multivitamin with Iron; Dietary Supplement: Chewable Calcium; Dietary Supplement: Quick Dissolve B12

INTERVENTIONS:
Dietary Supplement: Chewable Multivitamin with Iron — Take daily: Chewable Multivitamin with Iron. The chewable vitamins, vitamin chew, or vitamin rapid/quick-melts can be consumed after surgery when cleared by the surgeon.
  Other Names: Oral Vitamin Supplementation
  Arms: Oral vitamins
Dietary Supplement: PatchMD Vitamin D3/Calcium Patch — Wear daily: PatchMD Vitamin D3/Calcium patch. The patch can be worn immediately after surgery in order to prevent deficiencies, and we hope to show that this supplementation method can also promote lean muscle mass retention. In addition, due to the malabsorptive properties of bariatric surgery, we hope to show that patients will be more likely to completely absorb the micronutrient via transdermal application than through oral intake.
  Other Names: Transdermal Vitamin Supplementation
  Arms: Topical vitamin patch
Dietary Supplement: PatchMD Multivitamin Patch — Wear daily: PatchMD Multivitamin patch. The patch can be worn immediately after surgery in order to prevent deficiencies, and we hope to show that this supplementation method can also promote lean muscle mass retention. In addition, due to the malabsorptive properties of bariatric surgery, we hope to show that patients will be more likely to completely absorb the micronutrient via transdermal application than through oral intake.
  Other Names: Transdermal Vitamin Supplementation
  Arms: Topical vitamin patch
Dietary Supplement: PatchMD B12 Energy Plus Patch — Wear daily: PatchMD B12 Energy Plus patch. The patch can be worn immediately after surgery in order to prevent deficiencies, and we hope to show that this supplementation method can also promote lean muscle mass retention. In addition, due to the malabsorptive properties of bariatric surgery, we hope to show that patients will be more likely to completely absorb the micronutrient via transdermal application than through oral intake.
  Other Names: Transdermal Vitamin Supplementation
  Arms: Topical vitamin patch
Dietary Supplement: Chewable Calcium — Take daily: Chewable Calcium. The chewable vitamins, vitamin chew, or vitamin rapid/quick-melts can be consumed after surgery when cleared by the surgeon.
  Other Names: Oral Vitamin Supplementation
  Arms: Oral vitamins
Dietary Supplement: Quick Dissolve B12 — Take daily: Quick Dissolve B12. The chewable vitamins, vitamin chew, or vitamin rapid/quick-melts can be consumed after surgery when cleared by the surgeon.
  Other Names: Oral Vitamin Supplementation
  Arms: Oral vitamins

SUMMARY:
The objectives in this study are to provide information on the efficacy of transdermal supplement patches on treating nutrient malabsorption and deficiency in post-op bariatric patients, and to determine short-term body composition, HbA1c and fasting plasma glucose outcomes for patients after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients currently approved for vertical sleeve or gastric bypass bariatric surgery
* female patients should not be pregnant or plan to become pregnant

Exclusion Criteria:

* metal objects in the body
* current weight greater than 600lbs
* previous bariatric (revision) surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Fasting Blood Glucose | 3 months
  Glucose (mg/dL)
Calcium Blood Value | 3 months
  Calcium (mg/dL)
Iron Blood Value | 3 months
  Ferritin (ng/mL)
Vitamin B12 Blood Value | 3 months
  B12 (pg/mL)
Vitamin D Blood Value | 3 months
  Vitamin D, 25-Hydroxy (pg/mL)
HbA1c Blood Value | 3 months
  Hemoglobin A1c (%)
Fat Mass Measurement | 3 months
  Fat Mass (kg) via Tanita scale measurements
Fat Free Mass Measurement | 3 months
  Fat Free Mass (kg) via Tanita scale measurements
Weight Measurement | 3 months
  Weight (kg) via Tanita scale measurements
Waist Circumference | 3 months
  Waist circumference (cm)
Hip Circumference | 3 months
  Hip circumference (cm)

SECONDARY OUTCOMES:
Height | 3 months
  Statiometer measurement (cm)
Total Body Water | 3 months
  Total body water (kg) via Tanita scale measurements

CONTACTS AND LOCATIONS:
Overall Officials: Bonny Burns-Whitmore, DrPH, RD, Study Director — Cal Poly Pomona; David M Oliak, MD, Study Chair — Oliak Center for Weight Loss
Locations (1):
- Oliak Center for Weight Loss, Brea, California, United States

IPD SHARING:
Plan to Share IPD: No